CLINICAL TRIAL: NCT04978948
Title: Study of STIM1 Membrane Expression During Autoimmune Diseases
Brief Title: Study of STIM1 Membrane Expression
Acronym: STIMEX
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: STIMEX - 29BRC21.0025
Record Dates: First submitted 2021-05-04; First posted 2021-07-27 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Autoimmune Diseases
Keywords: autoimmune diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 venous blood samples/patient or 9 venous blood samples/patient for patients suffering from disease for which an increase in the membrane expression of STIM1 has been identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (18):
- Myasthénie: Blood samples will be collected
- Myopathie inflammatoire (Myosite): Blood samples will be collected
- Neuropathie autoimmune: Blood samples will be collected
- Néphropathies autoimmunes: Blood samples will be collected
- Hépatite auto-immune: Blood samples will be collected
- Pancréatite auto-immune: Blood samples will be collected
- Purpura Thrombopénique Immunologique: Blood samples will be collected
- Dermatose bulleuse: Blood samples will be collected
- Thyroïdite autoimmune: Blood samples will be collected
- Sclérose en plaque: Blood samples will be collected
- Sclérose latérale amyotrophique: Blood samples will be collected
- Polyarthrite Rhumatoïde: Blood samples will be collected
- Spondylarthrite axiale: Blood samples will be collected
- controls: Patients without autoimune desease* Blood samples will be collected
- Lichen plan buccal auto-immun (LPB): Blood samples will be collected
- lichen plan buccal allo-immun liée à une GvHD (" Graft versus Host Disease "): Blood samples will be collected
- Lupus érythémateux systémique: Blood samples will be collected
- Sclérodermie: Blood samples will be collected

SUMMARY:
The aim of this study is to determine the expression of STIM1 in the plasma membrane of lymphocytes from patients suffering from different autoimmune diseases in order to identify new pathologies of interest presenting an over-expression of STIM1PM.

This would allow to initiate, following this study, research and development programs on the use of anti-STIM1 antibodies in these identified autoimmune diseases of interest.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the autoimmune diseases

Exclusion Criteria:

* Treatment with rituximab in the previous 12 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 years old. Diagnosis of one of the autoimmune diseases of interest according to the commonly accepted classification criteria for each disease, regardless of the level of disease activity.
Sampling Method: Non-Probability Sample
Enrollment: 670 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
level of STIM1-PM | Day 0
  Membrane expression level of STIM1-PM on the surface of immune cells, measured by flow cytometry

SECONDARY OUTCOMES:
correlation between STIM1 expression and Clinical Score | Day 0
  Study of correlation between STIM1 expression on different cells and clinical scores of different autoimmune diseases or treatments received

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHRU de Brest - Service de rhumatologie, Brest, Brest
  - Centre Hospitalier des Pays de Morlaix, Morlaix, Brittany Region
  - Centre Hospitalier de Quimper, Quimper, Brittany Region
  - CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning two years and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.